CLINICAL TRIAL: NCT05632809
Title: REStoring lymphoCytes Using NKTR-255* After chemoradiothErapy in Solid Tumors (RESCUE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0925; NCI-2022-09970 (Other: NCI CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — NKTR-255; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NKTR-255 combination (Durvalumab) (Experimental): Participants will receive vein over about 30 minutes. Participants receive the first dose within 72 hours (3 days) after you complete CRT and the second dose at 3 weeks after you complete CRT. Then, you will receive NKTR-255 one (1) time every 4 weeks after that for up to 1 year.
  Durvalumab Participants will receive durvalumab by vein over about 30 minutes. You will receive the first dose at 3 weeks after you complete CRT therapy. Then, you will receive durvalumab one (1) time every 4 weeks after that for up to 1 year
  Interventions: Drug: NKTR-255; Drug: Durvalumab

INTERVENTIONS:
Drug: NKTR-255 — Given by IV (vein)
Drug: Durvalumab — Given by IV (vein)

SUMMARY:
To learn about the effects of the investigational drug NKTR-255 in combination with the standard drug durvalumab on locally advanced NSCLC when given after CRT.

DETAILED DESCRIPTION:
Primary Objectives:

1. Estimate the level of lymphocyte restoration after administration of NKTR-255 concurrently with durvalumab after chemoradiation. Absolute lymphocyte will be obtained along with changes in levels of NK cells, CD4 T cells, CD8 T cells, and B cells from baseline.
2. Monitor the safety of NKTR-255, which includes treatment related grade 3+ radiation pneumonitis

Secondary Objectives:

1. Estimate the Progression-free survival time distribution
2. Estimate the Overall survival time distribution

Exploratory objectives:

1. Characterize pharmacokinetics of NKTR-255 and assess immunogenicity of NKTR-255
2. Characterize pharmacodynamic effects and changes in activation markers and proliferation of NK and CD8 T cells, and cytokine levels after administration of NKTR-255 in combination with Durvalumab
3. Assess the correlation between ctDNA and efficacy measurements

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Histologic diagnosis of non-small cell lung cancer
3. Written consent obtained before initiation of any study-related procedures
4. Definitive cancer treatment intent
5. Absence of concurrent malignancies at other sites, except low risk prostate cancer and basal cell of the skin. Participants with prior cancers should not be receiving active cancer treatment within the past 3 months. Cancer survivors who have undergone potentially curative therapy for a prior malignancy who have no evidence of that disease for 1 year and who are deemed at low risk for recurrence are eligible for the study.
6. Adequate liver (AST, ALT, Alk Phos, and Tbili <2 fold upper limit) and kidney function (Cr < 2.5 limit of normal and Cr clearance >30)
7. ECOG 0-2

Exclusion Criteria:

Subjects are to be excluded from the study if any of the following conditions apply:

1. HIV infection, cellular immune deficiencies, hypogammaglobulinemia or dysgammaglobulinemia, or hereditary or congenital immunodeficiencies
2. Prior diagnosis of hepatitis B or C (unless anti-hepatitis C therapy has produced a sustained virologic response);
3. History of clinically significant autoimmune disease, Crohn's disease, ulcerative colitis, or inflammatory disease.
4. Serious concomitant disorder, including active systemic infection requiring treatment, as judged by the Investigator.
5. Known or suspected hypersensitivity to any component of the investigational product
6. Recurrent radiation to the treatment site
7. Prior major surgery within 4 weeks of enrollment from which the patient has not recovered
8. Other condition or prior therapy that, in the opinion of the Investigator, compromises the subject's welfare or may confound study results
9. Previous enrollment in this study
10. Pregnancy: a female subject defined as a WOCBP who has a positive urine pregnancy test (e.g. within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Prior exposure to any anti-PD-1 or anti-PD-L1 antibody.
12. Patients must be capable of understanding and providing a written informed consent.
13. Patients with leukemias or lymphomas with T cell/histiocyte or NK cell rich component(s) and other variants not otherwise specified that contain high numbers of T or NK cells.
14. Evidence of clinically significant interstitial lung disease or active noninfectious pneumonitis during the course of chemoradiation that is unresolved to ≤ grade 1.
15. Patients with grade 4 toxicities during chemoradiation not resolved to grade ≤ 1 by the end of chemoradiation.
16. Prior exposure to IL-2 or IL-5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival time distribution | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org